CLINICAL TRIAL: NCT04863690
Title: Assessing the Effects of the Muse Sleep Intervention on Sleep
Acronym: MuseSleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: InteraXon, Inc. (Industry); Cambridge Brain Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 118355
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mediation; Coaching
Keywords: Meditation; Sleep; Cognition
MeSH Terms: conditions — Negotiating | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep Intervention System - No Coaching (Experimental): Participants will be asked to use either the Muse Mind Meditation, Muse Sleep Journeys, Go to Sleep Soundscapes or Go to Sleep Guidance each evening as part of their bedtime routine to help them prepare to sleep. In addition, participants may use any part of the Muse App (Mind, Heart, Breath, Body, Guided or Go to Sleep meditations), as often as they like to help them fall asleep, go back to sleep, or as a meditation practice during the daytime. All Participants will also be asked to do the Muse Mind meditation for a minimum of 5 minutes per day, a minimum of 5 days per week, for 6 weeks.
  Interventions: Behavioral: Meditation
- Sleep Intervention System - Plus Digital Coaching (Experimental): The procedure will be identical to Group 1 above, but in addition, all participants will also work through the content in the Muse S Sleep Coaching course, and implement the sleep hygiene and habit changes recommended through the course that they find reasonable and effective for their situation.
  Interventions: Behavioral: Meditation; Behavioral: Digital Coaching
- Sleep Intervention System - Plus Digital Coaching plus Human Coaching (Experimental): The procedure will be identical to Group 2 above, but in addition, all participants will be asked to join regular online coaching sessions. Participants will be divided into 9 cohorts of 10 people per cohort. Each cohort will be offered group coaching once per week. Coaches will be versed in Mindfulness, and how to use Muse and how to support sleep. Coaching will take place virtually using Interaxon's Zoom account. Throughout the coaching, all participants will be referred to via their first names or their anonymized login names. In addition, for any challenges that arise, participants will have unlimited access to Muse Customer Care via phone, email, and video where appropriate during normal business hours.
  Interventions: Behavioral: Meditation; Behavioral: Digital Coaching; Behavioral: Digital Coaching plus Human Coaching
- Control (No Intervention): The participants in the control group will receive a Muse Device, which they will be free to keep at the end of the study. They will be asked not to open and/or use the Muse device until the entire study is complete. On day 1 of the Study, they will complete the Cambridge Brain Sciences online cognitive assessment battery), plus a longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and (depending on group), sleep quality. At the completion of the study controls will be offered optional, free group coaching sessions if they complete the study requirements.

INTERVENTIONS:
Behavioral: Meditation — Participants will be asked to use either the Muse Mind Meditation, Muse Sleep Journeys, Go to Sleep Soundscapes or Go to Sleep Guidance each evening as part of their bedtime routine to help them prepare to sleep. In addition, participants may use any part of the Muse App (Mind, Heart, Breath, Body, Guided or Go to Sleep meditations, as often as they like to help them fall asleep, go back to sleep, or as a meditation practice during the daytime. All Participants will also be asked to do the Muse Mind meditation for a minimum of 5 minutes per day, a minimum of 5 days per week, for 6 weeks. If they also wish to use the Muse system more frequently (day or night), they will be encouraged to do so and will be able to choose between several styles of available meditation (Mind, Heart, Breath, Body, Guided or Go to Sleep meditations). Participants will be asked to also wear their Muse device while they sleep, as often as they like in order to track their sleep.
  Arms: Sleep Intervention System - No Coaching; Sleep Intervention System - Plus Digital Coaching; Sleep Intervention System - Plus Digital Coaching plus Human Coaching
Behavioral: Digital Coaching — All participants will work through the content in the Muse S Sleep Coaching course, and implement the sleep hygiene and habit changes recommended through the course that they find reasonable and effective for their situation.
  Arms: Sleep Intervention System - Plus Digital Coaching; Sleep Intervention System - Plus Digital Coaching plus Human Coaching
Behavioral: Digital Coaching plus Human Coaching — All participants will work through the content in the Muse S Sleep Coaching course, and implement the sleep hygiene and habit changes recommended through the course that they find reasonable and effective for their situation. All participants will also be asked to join regular online coaching sessions. Participants will be divided into 9 cohorts of 10 people per cohort. Each cohort will be offered group coaching once per week. Coaches will be versed in Mindfulness, and how to use Muse and how to support sleep. Coaching will take place virtually using Interaxon's Zoom account.
  Arms: Sleep Intervention System - Plus Digital Coaching plus Human Coaching

SUMMARY:
In this study, we will examine whether use of the Sleep Intervention protocol marketed by Interaxon (the 'Muse'), leads to improvements in sleep quality (e.g. decreased latency to sleep, improved sleep duration), as well as knock-on improvements on measures of mindfulness, improvement in quality of life scores, reduction in perceived stress levels, anxiety, improvements in cognitive performance, improvement in markers relevant for safety, and increased success in the workplace in healthy participants.

DETAILED DESCRIPTION:
We all sleep, hopefully, every single day. Regular and sufficient sleep helps maintain numerous aspects of physical and mental health, but countless ordinary life circumstances, such as parenthood, demanding professions, studying, illness, or lifestyle choices often prevent people from getting a full night's sleep. In fact, in a recent US health survey of approximately 250000 people, 29.2% of respondents reported getting less than an average of 6 hours of sleep per night. Individuals who sleep this little on a day-to-day basis are considered to be experiencing chronic partial sleep deprivation (SD) (also known as sleep restriction), which, in a laboratory setting, has been associated with impaired physiological and cognitive functioning. It has been estimated that the productivity lost annually due to chronic partial SD costs an estimated $21.4 billion in Canada alone.

Interaxon markets a non-invasive head-worn device EEG biofeedback device ('Muse') to encourage and aid effective meditation and sleep. This device has been previously shown to improve workplace wellness, fatigue and quality of life, and performance on Stroop Task. It has also been shown to improve physiological markers associated with improved relaxation and cognition. Muse has been shown to have EEG signal comparable to a clinical grade EEG.

What is not known, is whether use of the Muse device can actually improve sleep quality and if so, in what ways. Thus far, some reports have suggested that the Muse Meditation device can improve relaxation, but a comprehensive evaluation of sleep has not been undertaken in a relatively large sample of healthy volunteers.

In this study, we will examine whether use of the Muse Sleep Intervention by healthy participants, leads to improvements in sleep quality (e.g. decreased latency to sleep, improved sleep duration), as well as knock-on improvements on measures of mindfulness, improvement in quality of life scores, reduction in perceived stress levels, anxiety, improvements in cognitive performance, improvement in markers relevant for safety, and increased success in the workplace. We will examine whether these changes are associated with changes in heart rhythm as measured by the Muse on board PPG sensor.

360 participants working in a large engineering firm, Hatch, will use the Muse Sleep Intervention to meditate before sleep over the course of 6 weeks.

The participants will be randomly divided into 4 groups with 90 participants in each group (see below).

Group 1 will use the Muse Sleep Intervention system with no coaching.

Group 2 will use the Muse Sleep Intervention system with digital coaching.

Group 3 will use the Muse Sleep Intervention system with digital coaching and additional human group online coaching.

Group 4 will be a control group and will not use any of the Muse meditation systems.

On day 1 of the Study, all participants will complete the Cambridge Brain Sciences online cognitive assessment battery, plus a longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and sleep quality. They will then begin the 6-week study according to their following Group assignments:

Group 1: Sleep Intervention System - No Coaching Participants will join a 1.5-hour virtual onboarding session where they will be trained on how to use the Muse S device and will complete their first Muse session. Participants will be asked to use either the Muse Mind Meditation, Muse Sleep Journeys, Go to Sleep Soundscapes or Go to Sleep Guidance each evening as part of their bedtime routine to help them prepare to sleep. In addition, participants may use any part of the Muse App (Mind, Heart, Breath, Body, Guided or Go to Sleep meditations), as often as they like to help them fall asleep, go back to sleep, or as a meditation practice during the daytime. All Participants will also be asked to do the Muse Mind meditation for a minimum of 5 minutes per day, a minimum of 5 days per week, for 6 weeks. If they also wish to use the Muse system more frequently (day or night), they will be encouraged to do so and will be able to choose between several styles of available meditation (Mind, Heart, Breath, Body, Guided or Go to Sleep meditations). Participants will be asked to also wear their Muse device while they sleep, as often as they like in order to track their sleep. Participants will have unlimited access to Muse Customer Care via phone, email, and video where appropriate during normal business hours.

Group 2: Sleep Intervention System - Plus Digital Coaching The procedure will be identical to Group 1 above, but in addition, all participants will also work through the content in the Muse S Sleep Coaching course, and implement the sleep hygiene and habit changes recommended through the course that they find reasonable and effective for their situation.

Group 3: Sleep Intervention System - Plus Digital Coaching plus Human Coaching. The procedure will be identical to Group 2 above, but in addition, all participants will be asked to join regular online coaching sessions. Participants will be divided into 9 cohorts of 10 people per cohort. Each cohort will be offered group coaching once per week. Coaches will be versed in Mindfulness, and how to use Muse and how to support sleep. Coaching will take place virtually using Interaxon's Zoom account.

Group 4: Controls The participants in the control group will receive a Muse Device, which they will be free to keep at the end of the study. They will be asked not to open and/or use the Muse device until the entire study is complete. On day 1 of the Study, they will complete the Cambridge Brain Sciences online cognitive assessment battery, plus a longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and (depending on group), sleep quality.

At the end of Week 6 (at the completion of the main study period), all participants will be reassessed using the Cambridge Brain Sciences online cognitive assessment battery, and the longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and sleep quality.

All participants will also complete a brief debriefing questionnaire at the end of Week 6, reporting their experiences about the study.

They will again be assessed using the Cambridge Brain Sciences online cognitive assessment battery, and the longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and sleep quality at the end of Week 12 (6 weeks after completing the main study period).

ELIGIBILITY:
Inclusion Criteria:

The study will be open to all Hatch employees in Canada. Hatch is a large engineering firm in Canada. Hatch currently has 4406 Canadian employees and therefore our sample size represents approximately 10% of the population.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Sleep Scores | 12 weeks
  The primary outcome will be scores on the Sleep Questionnaire. This questionnaire includes the Pittsburgh Sleep Quality Index which is the most widely accepted and validated self-report method for assessing changes in sleeping patterns.

SECONDARY OUTCOMES:
Score on the Cambridge Brain Sciences | 12 weeks
  Secondary outcome measures will be score on the Cambridge Brain Sciences (CBS) cognitive battery. The CBS battery assesses aspects of memory, attention, planning, and reasoning, using a web-based interface that can be self-administered at home through any internet browser.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian M Owen, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Canada

IPD SHARING:
Plan to Share IPD: No